CLINICAL TRIAL: NCT04131686
Title: A Cluster-randomized, Open, Prospective, Observational Study to Evaluate the Treatment Effectiveness and Safety of N-acetylcysteine(NAC) Inhalation Compared With Standard Treatment in Patients With Symptomatic Acute Rhinosinusitis
Brief Title: NAC Inhalation in the Treatment Of Symptomatic acuTe rhinosinUSitis
Acronym: NOTUS
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-NAC-OS-401
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Acute Rhinosinusitis; Recurrent Acute Rhinosinusitis; Chronic Rhinosinusitis
Keywords: rhinosinusitis; N-acetylcysteine
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control sites: Group of patients receiving standard treatment for symptomatic acute rhinosinusitis
- Test sites: Group of patients receiving NAC inhalation in addition to standard treatment for symptomatic acute rhinosinusitis

SUMMARY:
N-acetylcysteine (NAC), known to have mucolytic and antioxidant effects, is widely used to treat respiratory diseases and manage post-surgery pulmonary complications. It is also administered as a treatment for acetaminophen addiction and a preventive measure for contrast-induced nephropathy (CIN). While NAC inhalation is commonly used for mucolytic purpose for various respiratory disease because it has relatively less side effects compared to oral or injection administrations, it is more used as a part of allopathy than as a major therapy. As a result, there is neither enough relevant clinical data nor specific reference in treatment guidelines. Therefore, this study aims to evaluate the overall treatment effectiveness and safety of NAC inhalation compared with standard treatment, and to perform follow-up observations on administration cases, patient characteristics, and adverse events of NAC inhalation used in real clinical settings.

DETAILED DESCRIPTION:
Study Methodology :

12 medical institutions in Korea that meet the inclusion criteria are cluster-randomized (test sites : control sites =1:1). Information about randomization is disclosed to both investigators and subjects. This means both study center investigators and subjects will be aware of the purpose of this study as well as the result of randomization (whether the subjects will receive NAC inhalation or not) from the beginning of the study.

Investigators shall obtain voluntary consent for participation in this research from patients who visit their medical institutions with symptomatic acute rhinosinusitis within the study duration. Patients who provided a written consent for the use of their personal information and who satisfy inclusion/exclusion criteria will be given a study enrollment number and available data on these patients will be collected among the predefined study relevant data in the case reports until Day 14 (±3 days) from the starting day of treatment.

Statistical Analysis Methods (Analysis of primary endpoints) :

Obtain descriptive statistics (average, standard deviation, median, minimum, quartile, and maximum) for the change in the total score of the investigator's symptomatic severity assessment by treatment group on Day 14 compared with each time point and baseline (Day 0). Paired t-test shall be used to check intra-group change difference and Two sample t-test shall be used to check inter-group change difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients are explained about the study objectives and methodologies, and shall express their consent by signing a written agreement for the use of their personal information.
* Male and female patients who are ≥ 18 years old.
* Symptomatic acute rhinosinusitis patients whose symptoms have been present for more than 1 week and less than 12 weeks; recurrent acute rhinosinusitis patients (acute rhinosinusitis relapsed 3 times or more within 6 months, sub-clinical symptoms between the relapses); or, symptomatic acute-on-chronic (12 weeks or more) rhinosinusitis patients. [Patients display 2 or more symptoms that imply rhinosinusitis infection. The displayed symptoms should include at least one or more cardinal symptoms (nasal congestion or nasal/postnasal discharge).]
* The total score of the investigator's symptomatic severity assessment for a patient is 4 or above, and four symptomatic aspects (nasal congestion, nasal/postnasal discharge, facial pain/sense of facial pressure, reduction/loss of smell) are rated in four categories (0=no symptom, 1=mild, 2=moderate, 3=severe).
* Patients have anterior rhinoscopy or nasal endoscopy results, and one or more of the following are observed: Redness, Edema or mucosal obstruction(mostly in the middle nasal), Mucopurulent discharge(mostly in the middle nasal), Nasal polyps

Exclusion Criteria:

* Patients with rhinosinusitis of dental origin.
* Patients with a known chronic pulmonary symptoms including bronchial asthma and chronic bronchitis.
* Patients with nasal obstruction to the extent that drug administration is difficult.
* Patients who have received endoscopic sinus surgery within the last 3 months.
* Patients who have shown hypersensitivity or are likely to show hypersensitivity to N-acetylcysteine inhalation components (for the test sites)
* Pregnant or breast-feeding patients.
* Patients who are currently participating in other clinical trials (clinical trials for drugs or medical devices) or are planning to participate in other clinical trials during the duration of this study.
* Patients who are not suitable for study participation upon the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic acute rhinosinusitis (including recurrent acute rhinosinusitis and symptomatic acute-on-chronic rhinosinusitis).
  Approximately 300 subjects (Re-enrollment is not allowed.)
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: hospitals (sites)
Period: Overall Study
Arm/Group | Control Sites | Test Sites
Started | 146; 6 hospitals (sites) | 148; 6 hospitals (sites)
Completed | 138; 6 hospitals (sites) | 143; 6 hospitals (sites)
Not Completed | 8; 0 hospitals (sites) | 5; 0 hospitals (sites)

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Sites | Test Sites | Total
Number analyzed (Participants) | 138 | 143 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.69 (15.38) | 50.45 (15.20) | 51.55 (15.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 68 | 146
  Male | 60 | 75 | 135
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.14 (3.61) | 24.06 (3.36) | 24.11 (3.50)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total Score of the Investigator's Symptomatic Severity Assessment (Day 0, Day 14)
Description: Assessed symptoms: nasal congestion, nasal/postnasal discharge, facial pain/sense of facial pressure, reduction/loss of smell are rated in four categories [0=no symptom, 1=mild, 2=moderate, 3=severe] The total score is sum of the investigator's symptomatic assessment scores (on nasal congestion, nasal/postnasal discharge, facial pain/sense of facial pressure, and reduction/loss of smell); the maximum total score is 12 and minimum total score is 0
Time Frame: Day 0(enrollment) and Day 14 after treatment for rhinosinusitis
Population: Subject with investigator's symptomatic severity assessment was collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Sites | Test Sites
Number analyzed (Participants) | 135 | 137
score on a scale | -4.37 (2.04) | -3.56 (1.74)

ADVERSE EVENTS:
Time Frame: 14days
Description: Adverse drug reaction related to NAC inhalation was collected in the test sites and serious adverse event was collected in the whole study sites.
Arm/Group | Control Sites | Test Sites
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/143
Other Adverse Events (participants affected / at risk) | 0/138 | 7/143
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Sites (N=138) | Test Sites (N=143)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT04131686/Prot_SAP_000.pdf